CLINICAL TRIAL: NCT04957186
Title: Development of a Multidisciplinary Care Pathway With Postoperative Follow-up Via Electronic Patient Reported Outcomes (ePRO) of Complications of Breast Cancer Surgery to Optimise Patients' Quality of Life.
Brief Title: Personalized Follow-up After Breast Cancer Surgery Via Electronic Patient Reported Outcomes
Acronym: BEAUTIFY-2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Prix Ruban Rose/2021/FF-01
Record Dates: First submitted 2021-06-22; First posted 2021-07-12 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Breast Cancer
Keywords: Patient Reported Outcomes; Mastectomy; Postoperative Complications; Quality of Life; Breast Cancer
MeSH Terms: conditions — Breast Neoplasms; Postoperative Complications

STUDY DESIGN:
Intervention Model Description: There will be two groups in this study : one "Focus group" consisting of 10 patients who have undergone breast cancer surgery (tumorectomy, mastectomy, lymph node dissection), and one group of 10 caregivers consisting of 3 surgeons, 3 algologists, 3 oncologists and one study coordinator.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient Focus Group (Active Comparator): Group consisting of 10 patients who have undergone breast cancer surgery (tumorectomy, mastectomy, lymph node dissection).
  Interventions: Other: Collection of postoperative information
- Caregiver Focus Group (Active Comparator): Group consisting of 10 caregivers composed of 3 surgeons, 3 algologists, 3 oncologists and one study coordinator.
  Interventions: Other: Analysis of postoperative information collected from patients

INTERVENTIONS:
Other: Collection of postoperative information — The EORTC BR45 questionnaire will be used to gather information from patients regarding possible post-operative complications recorded via electronic patient-reported outcomes (pain, swelling, hypersensitivity etc.) as well as via the interviews with the state-registered coordinating nurse.
  Arms: Patient Focus Group
Other: Analysis of postoperative information collected from patients — All post-operative complications recorded via electronic patient-reported outcomes (pain, swelling, hypersensitivity etc.) as well as via the interviews with the state-registered coordinating nurse will be analyzed with the aim of proposing an appropriate care pathway.
  Arms: Caregiver Focus Group

SUMMARY:
Based on one focus group of caregivers and one group of patients treated by surgery for breast cancer this study is an attempt to identify the specific needs of this population and then develop the BEAUTIFY care pathway.This study aims to build a new multidisciplinary care pathway (BEAUTIFY = BrEast cAncer qUaliTy of lIfe aFter surgerY) with post-operative follow-up via electronic patient-reported outcomes of breast cancer surgery complications in order to optimize the quality of life of patients.

DETAILED DESCRIPTION:
This study aims to build a new multidisciplinary care pathway (BEAUTIFY = BrEast cAncer qUaliTy of lIfe aFter surgerY) with post-operative follow-up via electronic patient-reported outcomes of breast cancer surgery complications in order to optimise the quality of life of patients.

The study will use focus groups of caregivers and patients treated by surgery for breast cancer to identify the specific needs of this population and then develop the BEAUTIFY care pathway.

In oncology, the monitoring of symptoms and treatment toxicities by caregivers is most often done through hetero-assessments. However, caregivers tend to underestimate them in relation to what the patient is experiencing. The discrepancy between the measures of side-effects recorded by the doctor's and patient's measures of side effects has indeed been demonstrated many times. For the patient's own view of his or her symptoms, health symptoms, health status, or quality of life (QoL), the (QoL), Patient Reported Outcomes (PRO) are increasingly used in oncology. They are defined as "any measure of the patient's health status reported directly by the patient, without interpretation by the physician or a third person". Several clinical trials have been conducted in recent years to assess the feasibility and value of collecting PROs in clinical routine in oncology, particularly through the use of electronic objects (ePROS). Improvements have been shown in the overall survival and QoL of patients followed by ePROS compared to conventionally followed patients, in patients on chemotherapy for metastatic cancer and in lung cancer surveillance.

Breast cancer surgery is responsible for specific acute (infection, haematoma, pain) and chronic (breast pain, axillary pain, arm pain, allodynia, paresthesia, retractile capsulitis of the shoulder post-mastectomy syndrome). Acute infections Post-operative infections may occur in 3 to 19% of 2020 RUBAN ROSE patients, especially after mastectomy. Chronic pain is reported in up to 70% of patients depending on the series. Post-mastectomy syndrome affects 20 to 50% of patients. These complications may be increased by radiotherapy. Many studies have shown that all of these chronic complications have a negative impact on the quality of life of patients and are responsible for depression and/or anxiety, sleep disorders and difficulties in returning to work.

Nevertheless, there are specific treatments (PEC) that can reduce these symptoms: physiotherapy, analgesic medication, analgesic patches, botulinum toxin injections, psychotherapy, etc. Several studies have shown that the earlier this treatment is undertaken, the lower the risk of complications.

It is therefore necessary to detect these complications as early as possible in order to manage them as quickly as possible. A close follow-up of specific symptoms of breast cancer surgery complications by ePRO could lead to earlier detection and management of these complications and thus improve patients' pain and quality of life (QoL).

We propose to develop an original care pathway focused on the collection of post-surgery complications in breast cancer via ePROs. The BEAUTIFY programme will be built by a committee of experts on the basis of reflections carried out within 2 focus groups: a group of 10 patients treated at Nîmes University Hospital for breast cancer; a group of caregivers from the University Hospitals of Nîmes, Montpellier and the ICM.

ELIGIBILITY:
Inclusion Criteria:

* Female adult patients recruited from the gynecological or medical oncology department at Nîmes University Hospital who have undergone breast cancer surgery at least 6 months previous to their inclusion in the study and recruited during their post-operative follow-up consultations.
* All patients must have given written informed consent.

Exclusion Criteria:

* Patients who have not undergone breast cancer surgery.
* Patients Under the age of 18.
* Patients who have not given written informed consent.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 20 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Specific needs of patients who have undergone breast cancer surgery : ePRO results | Up to 1 month following the end of radiotherapy treatment
  Electronic Patient Reported Outcomes (ePROs) will be used to record postoperative complications of these patients who have undergone breast cancer surgery. Patients will have to express themselves according to items 47 - 53 of the EORTC QLQ-BR45 questionnaire containing questions related to the previous Week. The patient must answer on a scale of 1 to 4 in which 1 = Not at All, 2 = A little, 3 = Quite a Bit and 4 = Very Much
Use of ePROs as a means of collecting post-surgical complications | Up to 1 month following the end of radiotherapy treatment
  Patients will be asked to give their appreciation of the use of Electronic Patient Reported Outcomes (ePROs) to record their postoperative complications: time taken, frequency and the type of interface used (ePRO or telephone)
Results of the interview with the nurse for collecting post-surgical complications | Up to 1 month following the end of radiotherapy treatment
  Patients will be asked to give their appreciation of the interview with the nurse to record their postoperative complications.
Actions desired in the event of an onset of complications in patients who have undergone breast cancer surgery. | Up to 1 month following the end of radiotherapy treatment
  Patients will be asked to express what actions they would like to be undertaken in the event of an onset of complications.
Degree of anxiety/reassurance of patients who have undergone breast cancer surgery. | Up to 1 month following the end of radiotherapy treatment
  Patients will be asked to express their degree of anxiety or reassurance following their breast cancer surgery according to a Lickert scale of 1 to 5 in which 1 = completely reassured, 2 = reassured, 3 = indifferent, 4 = anxious and 5 = extremely anxious.
Expectations of patients who have undergone breast cancer surgery. | Up to 1 month following the end of radiotherapy treatment
  Patients will be asked to express their expectations of the results of this information-gathering. These will be expressed on a Lickert scale of 1 to 5 in which 1 = not very hopeful, 2 = hopeful, 3 = indifferent, 4 = very hopeful, 5 = extremely hopeful.

CONTACTS AND LOCATIONS:
Locations (1):
- Nîmes University Hospital, Nîmes, Gard, France

REFERENCES:
- [Background] Di Maio M, Basch E, Bryce J, Perrone F. Patient-reported outcomes in the evaluation of toxicity of anticancer treatments. Nat Rev Clin Oncol. 2016 May;13(5):319-25. doi: 10.1038/nrclinonc.2015.222. Epub 2016 Jan 20. PMID 26787278
- [Background] Basch E, Deal AM, Dueck AC, Scher HI, Kris MG, Hudis C, Schrag D. Overall Survival Results of a Trial Assessing Patient-Reported Outcomes for Symptom Monitoring During Routine Cancer Treatment. JAMA. 2017 Jul 11;318(2):197-198. doi: 10.1001/jama.2017.7156. PMID 28586821
- [Background] Kitzinger J, Barbour RS.Developing Focus Group Research: Politics, Theory and Practice. SAGE 1999
- [Background] Hamood R, Hamood H, Merhasin I, Keinan-Boker L. Chronic pain and other symptoms among breast cancer survivors: prevalence, predictors, and effects on quality of life. Breast Cancer Res Treat. 2018 Jan;167(1):157-169. doi: 10.1007/s10549-017-4485-0. Epub 2017 Aug 31. PMID 28861642
- [Background] Montemurro F, Mittica G, Cagnazzo C, Longo V, Berchialla P, Solinas G, Culotta P, Martinello R, Foresto M, Gallizioli S, Calori A, Grasso B, Volpone C, Bertola G, Parola G, Tealdi G, Giuliano PL, Aglietta M, Ballari AM. Self-evaluation of Adjuvant Chemotherapy-Related Adverse Effects by Patients With Breast Cancer. JAMA Oncol. 2016 Apr;2(4):445-52. doi: 10.1001/jamaoncol.2015.4720. PMID 26720497
- [Background] Scaffidi M, Vulpiani MC, Vetrano M, Conforti F, Marchetti MR, Bonifacino A, Marchetti P, Saraceni VM, Ferretti A. Early rehabilitation reduces the onset of complications in the upper limb following breast cancer surgery. Eur J Phys Rehabil Med. 2012 Dec;48(4):601-11. Epub 2012 Apr 17. PMID 22510674